CLINICAL TRIAL: NCT00207298
Title: Phase III Open Label Trial for Use of [18F]-Fluoro-Deoxy-Glucose (18F-FDG) in Positron Emission Tomography Imaging in Oncology
Brief Title: 18F-fluorodeoxyglucose (18F-FDG) Positron Emission Tomography in Oncology
Status: Completed | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: R05-0076
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Brain Neoplasms; Lung Neoplasms; Lymphoma; Melanoma; Colorectal Neoplasms
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Lymphoma; Melanoma; Colorectal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Positron Emission Tomography — Each patient will receive an 18F-FDG PET/CT scan

SUMMARY:
Positron emission tomography (PET) is a nuclear medicine procedure based on the measurement of positron emission from radiolabelled tracer molecules. These radiotracers allow biologic processes to be measured and whole body images to be obtained which demonstrates sites of radiotracer accumulation. The most common radiotracer in use today is 18F-fluorodeoxyglucose (18F-FDG) which is a radiolabelled sugar (glucose) molecule. Imaging with 18F-FDG PET is used to determine sites of abnormal glucose metabolism and can be used to characterize and localize many types of tumours.

Cancer treatment and outcome depend largely on the accurate diagnosis and staging of disease. There is extensive data in the literature indicating the importance of FDG-PET imaging in accurately characterizing disease, as well as determining stage and sites of recurrent disease in many cancer types. For these indications, functional imaging with PET provides unique information which is not available from standard medical imaging modalities such as ultrasound, X-ray, computerized tomography (CT) or magnetic resonance imaging (MRI).

The objectives of this study are to document the safety and efficacy of 18F-FDG produced by the British Columbia Cancer Agency (BCCA) at its Tri-University Meson Facility (TRIUMF) production facility and to evaluate FDG-PET as a diagnostic and decision making tool in the management of oncology patients in British Columbia. With a population base of over 4 million people, standardized cancer treatment protocols, and evidence based guidelines for FDG-PET imaging, the BCCA is positioned to make an important contribution to defining the role of PET in the Canadian health care system.

DETAILED DESCRIPTION:
1.0 Background & Introduction

In general, diagnostic imaging can address two issues: structure and function. One can either view structures in the body and image anatomy using structural imaging modalities such as plain film radiography (X-ray), Computerized Tomography (CT) and Magnetic Resonance Imaging (MRI), or one can view chemical processes and image biochemistry and function using biochemical imaging modalities such as Planar and Single Photon Emission Computerized Tomography (SPECT) imaging and Positron Emission Tomography (PET). The strength of the biochemical imaging methods is in distinguishing tissues according to metabolism rather than structure.

18F-Fluorodeoxyglucose (FDG) is the most commonly used tracer for PET imaging; its use and safety are well established world wide. The 18F-FDG is injected intravenously and is transported from blood to tissues in a manner similar to glucose. It has been understood for over 50 years, that cancer cells, in general, have increased glucose uptake and anaerobic metabolism compared to normal tissues. Like glucose, FDG is taken up into cells through glucose transport proteins (GLUT) and then phosphorylated by hexokinase to FDG-6-phosphate. However, since FDG-6-phosphate is not a substrate for subsequent glucose metabolic pathways and has a very low membrane permeability, the FDG-6-phosphate becomes trapped in tissue in proportion to the rate of glycolysis. This accumulation of 18F-FDG-6-phosphate forms the basis of tumor metabolic imaging with PET.

2.0 Indications

Cancer treatment and outcome depend largely on the accurate diagnosis and staging of disease. There is extensive data in the literature indicating the importance of PET imaging in accurately characterizing disease, determining stage and sites of recurrent disease in many cancer types. For these indications, it is well documented in the literature that functional imaging with PET exceeds sensitivity, specificity and accuracy of conventional 3-D imaging modalities. The most widely cited reference for the efficacy of PET imaging is: A Tabulated Summary of the FDG PET Literature, published by Gambhir et al, JNM (2001) 42: 1S-93S. In this study the average FDG PET sensitivity and specificity across all oncology applications are estimated at 84% (based on 18,402 patient studies) and 88% (based on 14,264 patient studies), respectively. The average management change across all applications is estimated to be 30% (based on 5,062 patients). Data was obtained combining 419 total articles and abstracts on studies in which FDG PET was used. Various methods of analysis were applied to these data, which revealed only a small amount of variation in the ratio values. Specifically, the sensitivity of PET ranged from 84 - 87%, the specificity ranged from 88% - 93%, and the accuracy ranged from 87 - 90%.

In the United States, the Food and Drug Administration (FDA) has approved 18F-FDG for use in all cancer types. On January 28, 2005 the Centers for Medicare and Medicaid Services (CMS) announced that it would reimburse PET imaging studies when performed for almost all previously non-covered oncology indications. All previous PET coverage remained fully in effect, and initial staging of cervical cancer was added without conditions but coverage was expanded conditionally to include all cancers and non-covered indications except breast cancer diagnosis and regional lymph node staging.

(http://www.cms.hhs.gov/mcd/viewncd.asp?ncd_id=220.6.15&ncd_version=1&basket=ncd%3A220%2E6%2E15%3A1%3APET+%28FDG%29+for+All+Other+Cancer+Indications+Not+Previously+Specified)

The indication for performing this diagnostic imaging test is the need for non-invasive, functional assessment of patients suspected of having or previously diagnosed with:

* Lymphoma
* Colorectal cancer
* Breast cancer
* Esophageal cancer
* Head & neck cancer
* Melanoma
* Brain tumors
* Cervical cancer
* Testicular (Germ Cell) cancer
* Thyroid cancer
* Lung cancer
* Sarcoma

3.0 Study Objectives

Objectives of this study are to validate the safety of 18F-FDG produced by BCCA and to evaluate 18F-FDG PET as a decision making and diagnostic tool in the management of oncology patients in British Columbia. With a population base of over 4 million people, standardized cancer treatment protocols, and evidence-based guidelines for PET imaging, the BCCA is positioned to make an important contribution to defining the role of PET in the Canadian health care system.

4.0 Study Design

This will be a single cohort observational study design in which additional safety data will be collected from the first patient being scanned from each of the first three batches of 18F-FDG delivered to our clinical site. Data will be collected from referring physicians with respect to how the PET scan results affected patient management and results of the PET scan will be correlated with biopsy results when available. All subjects are informed of anticipated effects (none) and purpose of the injected substance. There is no intent to change the way this protocol is conducted or to in any way alter the effect or purpose of the injected tracer. Subjects are approached with respect to their willingness to participate in the proposed study based on clinical criteria and undergo a brief clinical assessment followed by scanning as outlined below.

5.0 Study Time-Frame

The B.C. Cancer Agency anticipates a start date in June 2005 and a potential completion date in August of 2015, at which time our on-site (Vancouver Cancer Centre) radiopharmacy and cyclotron will be operational. Ten years of data collection will provide meaningful numbers for analysis and support of an 18F-FDG New Drug Submission (NDS) to Health Canada.

6.0 Patient Population and Sample Size

A total of 40,000 patients will be entered into the study. This number is based on the anticipated number of PET scan referrals based on the criteria for study inclusion outlined below and our clinical capacity of 15 to 35 patients per day operating 220 days per year. This will be the only publicly funded PET program in the province of British Columbia. A sample size of 40,000 patients will allow the PET program in BC to operate until Phase B of the Functional Imaging Program is implemented and the BCCA is positioned to submit an NDS for 18F-FDG.

Assuming a response rate of 90% to the patient management survey and a change in patient management for 30% of the study participants, precision for the 95% confidence interval of the estimated proportion will be .013. Given the same response rate and change in patient management proportion, a tumour site with 100 patients will yield a precision of .089 for its 95% confidence interval.

A sensitivity (or specificity or accuracy) rate of 80% can be estimated for the full sample with a precision of .011 for its 95% confidence interval, or a precision of .080 for a sub-sample of 100.

Additional safety data will be collected from the first patient imaged from each of the first three batches of FDG delivered to our clinical site (N=3). The chemical structure of our product is identical to authentic FDG. We have performed a minimum of five consecutive 18F-FDG productions with all quality control passing and will have done many more in the course of this CTA review process. The safety record of FDG PET worldwide is undisputable and we expect the number of adverse events in our study to be zero. In addition to baseline assessment, these subjects will have their blood pressure, oxygen saturation, heart rate and temperature monitored every 15 minutes for 2 hours post-procedure. Patients will be questioned as to their general well-being after the scan. If there are concerns that the patients' health status has changed during or immediately following the scan, then a physician will provide a more detailed assessment. Each of these three patients will be followed up by telephone, usually the day after the scan to help insure there were no delayed effects. These whole body PET scan images will be reviewed independently by two Nuclear Medicine physicians to confirm an expected biodistribution of radioactivity. If a subject did experience a reaction post-injection that could not immediately be attributed to another condition or exposure, or if the biodistribution of FDG in normal tissue was altered and could not be explained on clinical grounds (eg. patient on G-CSF), the tracer would be re-examined and tested for impurities and pyrogens. The safety data collected from these three patients will verify that the FDG produced by the BCCA is behaving as expected.

Patients considered appropriate for participation in this protocol are drawn from a population made up of the following parameters:

* Patients are between the ages of 19 and 90 years, although exceptions to these numbers may be made depending on the individual's ability to understand, give assent/consent, and tolerate the procedure. Health Canada can expect a separate CTA submission from the BCCA within the next few months for FDG-PET indications in the pediatric oncology population.
* Patients are both female and male and of any race with no preference for any group over another.
* Patients are those who are suspected of having or who have been previously diagnosed with cancer and meet BCCA evidence-based guidelines for FDG-PET.

7.0 Inclusion Criteria

* Age 19 years or older.
* ECOG performance status 0 - 3.
* Able to provide written informed consent.
* Referred by a treating physician.
* Must meet BCCA Evidence-Based guidelines for FDG-PET in Oncology
* Patients must be able to tolerate the physical/logistical requirements of completing a PET scan including lying flat for up to 45 minutes and tolerating intravenous cannulation for injection.

8.0 Exclusion Criteria

* Patients' blood glucose > 11.1 mmol/L (200 mg/dL) measured by glucometer immediately prior to scan.
* Pregnancy.
* Patients unable to provide informed consent.
* Patients who are medically unstable eg. acute cardiac or respiratory distress, hypotensive
* Patients who exceed the safe weight limit of the PET/CT bed (204.5 kg) or who cannot fit through the PET/CT bore (diameter 70 cm).

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older.
* ECOG performance status 0 - 3.
* Able to provide written informed consent.
* Referred by a treating physician.
* Must meet BCCA evidence-based guidelines for FDG-PET in oncology
* Patients must be able to tolerate the physical/logistical requirements of completing a PET scan including lying flat for up to 45 minutes and tolerating intravenous cannulation for injection.

Exclusion Criteria:

* Patients' blood glucose > 11.1 mmol/L (200 mg/dL) measured by glucometer immediately prior to scan.
* Pregnancy
* Patients unable to provide informed consent.
* Patients who are medically unstable e.g. acute cardiac or respiratory distress or hypotensive
* Patients who exceed the safe weight limit of the PET/CT bed (204.5 kg) or who cannot fit through the PET/CT bore (diameter 70 cm).

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients in British Columbia who meet the eligibility requirements.
Sampling Method: Non-Probability Sample
Enrollment: 39242 (Actual)
Dates: Start 2005-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in management based on PET procedure | Up to 6 weeks

SECONDARY OUTCOMES:
Sensitivity of PET | Up to 6 weeks
Safety of 18F-FDG | Up to 24 hours after completion of PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Don C Wilson, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BCCA, Vancouver Centre, Vancouver, British Columbia, Canada

REFERENCES:
- See also: British Columbia Cancer Agency website — http://www.bccancer.bc.ca